CLINICAL TRIAL: NCT01557036
Title: Aneurysm Study of Pipeline in an Observational Registry
Acronym: ASPIRE
Status: Terminated | Type: Observational
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Other Study IDs: PED002
Record Dates: First submitted 2012-03-13; First posted 2012-03-19 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Brain Aneurysm
Keywords: Brain Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Aneurysms treated with Pipleline: Aneurysms treated with Pipleline. All patients independently treated according to the labeled indications for use with the Pipeline Embolization Device
  Interventions: Device: Pipeline Embolization Device

INTERVENTIONS:
Device: Pipeline Embolization Device — Aneurysms treated independent of study entry with the Pipeline Embolization Device. This is an observational, non-interventional study.
  Other Names: PED

SUMMARY:
The primary objective of this study is to further expand the body of clinical knowledge in patients undergoing Pipeline Embolization Device (Pipeline or PED) placement for intracranial aneurysms (IAs or ICAs) according to Pipeline's labeled indication.

ELIGIBILITY:
Inclusion Criteria:

(All sites, All countries)

1. At least 1 Pipeline placed for treatment of an ICA
2. Patient or patient's Legally Authorized Representative (LAR) has signed an IRB- or EC-approved informed consent form, if required
3. Patient is willing and able to comply with follow-up visits

United States: Additional Inclusion Criteria for subjects enrolled in the United States:

4US) Subjects who are age 22 or higher 5US) IA of at least 10 mm in maximum dimension along the internal carotid artery between the petrous and superior hypophyseal segments

Canada: Additional Inclusion Criteria for subjects enrolled in Canada:

4C) In Canada, the Pipeline™ Embolization Device is intended for use with or without embolic coils for the treatment of complex intracranial aneurysms that are not amenable to treatment with surgical clipping.

5C) Canadian licensing/approval is limited to devices that are between 3.25 mm and 5.00 mm in diameter.

France: Additional Inclusion Criteria for subjects enrolled in France:

4F) Unruptured IA, saccular or fusiform with an aneurysm sac diameter > 15mm and not treatable with other current therapies ( EVT with coils with or without assisting system (intracranial stent) or balloon remodeling, or surgery) due to its specific morphology.

5F) IA previously treated with unruptured recanalization of the aneurismal sac > 7 mm, not treatable with conservative treatment.

Exclusion Criteria: (based on contraindications PED IFU)

1. Active bacterial infection
2. A patient in whom dual antiplatelet therapy (aspirin and clopidogrel) is contraindicated
3. A patient who has not received dual antiplatelet agents prior to the procedure
4. Pre-existing stent is in place in the parent artery at the target aneurysm location
5. Angiography demonstrates inappropriate anatomy, e.g., severe pre-or post-aneurysm narrowing
6. Acutely ruptured aneurysm, defined as rupture of the target aneurysm Each site should refer to their country specific Instructions for Use/Approval(France) to determine final eligibility into the ASPIRe Registry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with an intracranial aneurysm meeting the labeled indication for the relevant geography.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Neurological Adverse Events following PED use | From Device placement until last follow up, for an average of 3 years of follow up for each subject enrolled
  The primary endpoint will consist of a composite of any/all of the events listed below.
  * Incidence of spontaneous rupture of Pipeline treated aneurysm
  * Incidence of other (non-aneurysmal) intracranial hemorrhage, ipsilateral and contralateral
  * Incidence of ischemic stroke
  * Incidence of symptomatic and asymptomatic parent artery stenosis
  * Incidence of permanent cranial neuropathy
  * Incidence of change in baseline neurologic signs/symptoms related to Pipeline treated ICA(s) at last assessment

CONTACTS AND LOCATIONS:
Locations (36):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Neurosurgical Associates, Phoenix, Arizona
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Radiology Imaging Associates / Colorado Neurological Institute, Englewood, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Neurointerventional Associates, P.A., St. Petersburg, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Neurosurgical Associates at Central Baptist, Lexington, Kentucky
  - Norton Neuroscience Institute, Louisville, Kentucky
  - Abbott Northwestern Hospital/Consulting Radiologists, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - St. Paul Radiology, Saint Paul, Minnesota
  - Washington University, St Louis, Missouri
  - University of Buffalo Neurosurgery, Buffalo General Hospital, Buffalo, New York
  - The State University of New York, Stony Brook, Stony Brook, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Luke's Episcopal Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Medical College Of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin
- Clínica La Sagrada Familia, Buenos Aires, Argentina
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Royal University Hospital, Saskatoon, Saskatchewan, Canada
- France (3):
  - Besançon University Hospital, Besançon
  - Hôpital Gui de Chauliac, Montpellier
  - Hôpital Maison Blanche - CHU, Reims
- Germany (2):
  - Alfried Krupp Krankenhaus, Essen
  - Klinikum Stuttgart, Stuttgart
- Italy (3):
  - Niguarda CA Granda Hospital of Milan, Milan
  - Fondazione Istituto Neurologico "Besta", Milan
  - Ospedale San Giovanni Bosco ASL Napoli 1 Centro, Napoli
- University Hospitals of Geneva (HUG), Geneva, Switzerland